CLINICAL TRIAL: NCT02047253
Title: A Phase 2 Trial of Carfilzomib for Metastatic Castration-resistant Prostate Cancer Following Chemotherapy and Androgen Pathway Inhibitors
Brief Title: Phase 2 Trial of Carfilzomib for Metastatic Castration-resistant Prostate Cancer Following Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Guru Sonpavde, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F130725012 (UAB 1336)
Record Dates: First submitted 2014-01-20; First posted 2014-01-28 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: carfilzomib; prostate cancer; PSA (prostate-specific antigen); CRPC (castration-resistant prostate cancer)
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic | interventions — carfilzomib; Dexamethasone; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib is administered twice-weekly on consecutive days (days 1, 2, 8, 9, 15, 16) as a 30-minute intravenous infusion for 3 weeks every 4 weeks (1 cycle) with dexamethasone given as pre-medication. The dose of carfilzomib is 20 mg/m2 on days 1 and 2 of cycle 1 and is then escalated in succeeding weeks and cycles to 56 mg/m2 if no dose limiting toxicities occur. Acyclovir is given orally at 400 mg twice daily during therapy but may be discontinued at some point. Therapy will continue until side effects become unacceptable, the disease progresses, or the doctor withdraws the patient.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Acyclovir

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be administered on days 1, 2, 8, 9, 15, 16 within each 4 week cycle.
  Other Names: Kyprolis
Drug: Dexamethasone — Administered prior to administration of Study drug
Drug: Acyclovir — Administered orally twice daily
  Other Names: Zovirax

SUMMARY:
This study will test how effective the drug, Carfilzomib, reduces progression of prostate cancer in patients who have previously received chemotherapy and androgen inhibitors. Carfilzomib is approved for multiple myeloma but is not approved for prostate cancer. Therefore, it is considered investigational. Other approved methods of treatment for metastatic prostate cancer have demonstrated only modest benefits. Novel and tolerable agents are necessary to make further gains and extend overall survival.

DETAILED DESCRIPTION:
First-line chemotherapy for metastatic castration-resistant prostate cancer (CRPC) combined with androgen inhibitors modestly extends overall survival. Carfilzomib is anticipated to enhance progression-free survival (PFS) as well as reduce pain and toxicities.

Proteasome inhibitors are promising agents used in the therapy of prostate cancer. Carfilzomib is a more potent and irreversible proteasome inhibitor than the frequently used proteasome inhibitor, Bortezomib. In Phase I trials Carfilzomib demonstrated substantial antitumor activity while exhibiting tolerable side effects.

Carfilzomib has been approved by the FDA for patients with multiple myeloma. The drug, however, is not approved for the use with CRPC patients. This trial will evaluate the tolerance and effectiveness of Carfilzomib in men with metastatic progressive CRPC following chemotherapy and androgen inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Metastatic disease
* Progressive disease (PSA, radiologic, symptomatic) following abiraterone acetate and/or Enzalutamide (prior sipuleucel-T and chemotherapy are allowed); PSA progression is defined as baseline increase followed by any PSA increase ≥1 week apart.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patients, even if surgically sterilized (i.e., status post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse if female partner of childbearing age.
* An elevated PSA level of >2ng/mL for patients progressing by PSA criteria is required (last confirmatory sample must be >2ng/mL)
* Currently on androgen ablation hormone therapy (a luteinizing hormone- releasing hormone (LHRH) agonist/antagonist or orchiectomy) with testosterone level <50ng/dL)
* Has an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 - 2
* Left ventricular ejection fraction (LVEF) ≥40% on 2-D transthoracic echocardiogram (ECHO); Multi-gated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
* ≥19 years of age
* Resolution of all acute toxic effects of prior chemotherapy or surgical procedures to NCI CTCAE Version 4.03 Grade <1, in the opinion of the treating physician.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patient has a platelet count of <100,000/mm3, or absolute neutrophil count of <1500/mm3 or Hemoglobin <8.0gm/dL
* Patient has a calculated or measured creatinine clearance of <30 milliliters (mL)/minute
* Patient has total bilirubin >2 x upper limit of normal (ULN), or aspartate aminotransferase (AST), alanine aminotransferase (ALT) >3.5 x ULN
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Before study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of: a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the breast; c) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
* Known HIV, hepatitis B and hepatitis C infection
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to randomization
* Prior treatment with bortezomib
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize Carfilzomib)
* Has received prior radiation to >50% of the bone marrow
* Has had significant bleeding/thrombosis in previous 4 weeks
* Has received treatment with radiation therapy, surgery, chemotherapy, or an investigational agent within 4 weeks prior to registration, (6 weeks for radiation therapy, radionuclides, nitrosoureas, or Mitomycin C) or who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Has evidence of uncontrolled Central Nervous System (CNS) involvement (previous radiation and off steroids is acceptable)
* Patients may not be receiving any other investigational agents
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection
* Is unable to comply with study requirements
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guru Sonpavde, MD, Principal Investigator — University of Alabama at Birmingham; Mansoor Saleh, MD, Study Chair — Georgia Cancer Specialists
Locations (4):
- United States (4):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cancer Life Center, Navicent Health, Macon, Georgia
  - University of Tulane, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: April 2014, Primary Completion Date: June 2017 and Study Completion Date: July 14, 2017. Recruitment location: University of Alabama at Birmingham (UAB) Comprehensive Cancer Center, Birmingham; Tulane University, New Orleans; Medical Center of Central Georgia, Macon, Georgia, Dana Farber Cancer Institute, Boston.
Period: Overall Study
Arm/Group | Carfilzomib
Started | 28
Completed | 20
Not Completed | 8
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The study will measure patient survival at 6 months but will continue to monitor overall survival as a secondary objective. The Kaplan-Meier method will be used.
Time Frame: Baseline through 6 months for evaluating all patients
Population: 8 patients did not complete treatment and were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 20
Participants | 1

2. Primary Outcome: Overall Survival
Description: Outcome measure was completed by using a count of participants.
Time Frame: From baseline through 36 months.
Population: 8 patients did not complete treatment and were lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 20
Participants | 11

3. Secondary Outcome: Number of Participants With Prostate-Specific Antigen (PSA) Changes
Description: PSA levels were collected at each visit on the day of treatment. Linear regression with PSA as the dependent variable and time as the dependent variable was performed.
Time Frame: Baseline through 36 months
Population: We were unable to collect blood specimen for PSA analysis for 1 patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 27
Participants | 3

4. Secondary Outcome: Number of Participants With Circulating Tumor Cell (CTC) Decline Over Three Time Points (Before Study Initiation, Day 1 of Cycles 2 and 4
Description: The CTC marker will be used to evaluate efficacy of response to treatment. CTC changes will include changes from unfavorable (less than or equal to 5/7.5 ml) to favorable and declines by >30%.
  Three collections: before study initiation, Day 1 of Cycles 2 and 4
Time Frame: Baseline through 36 months
Population: 1 patient did not have blood draw. 27 patients had blood draws for CTC enumeration across baseline, Cycle 2 day 1 and cycle 4 day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 27
Participants
  CTC decline | 3
  CTC increased or No change/decline in CTC levels | 24

5. Secondary Outcome: Assessment of Toxicities
Description: Hematologic and non-hematologic toxicities will be graded. The new international criteria proposed by the Response Evaluation Criteria In Solid Tumors (RECIST) will serve as the guideline.
  On Day 1 of each cycle (4 weeks) for the duration of treatment and then 30 days following the last treatment
Time Frame: Baseline through 36 months
Population: All serious adverse events and > grade 3 toxicities were reported for patients who received treatment with Carfilzomib
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 28
Participants
  Anemia (>= Grade 3 or 4) | 3
  Hypertension (>= Grade 3 or 4) | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 36 months.
Arm/Group | Carfilzomib
All-Cause Mortality (participants affected / at risk) | 6/28
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=28)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hypertension (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02047253/Prot_SAP_000.pdf